CLINICAL TRIAL: NCT05092906
Title: Randomized Controlled Study Evaluating The Contribution of a Hypnosis Intervention During a Lumbar Puncture in the Neurology Department.
Brief Title: Contribution of Hypnosis During a Lumbar Puncture.
Acronym: HYPNOPLUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 38RC20.357
Record Dates: First submitted 2021-09-16; First posted 2021-10-26 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Pain
Keywords: lumbar puncture; anxiety
MeSH Terms: conditions — Pain; Anxiety Disorders | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lumbar puncture with standard of care (Active Comparator)
  Interventions: Other: LP with standard of care
- Lumbar puncture with hypnosis add-on therapy (Experimental)
  Interventions: Other: LP with complementary hypnoanalgesia

INTERVENTIONS:
Other: LP with complementary hypnoanalgesia — The lumbar puncture technique will be identical to that of the group standard of care. Hypnosis will be performed by a health professional trained in this practice, in addition to the standard analgesic management.
  Arms: Lumbar puncture with hypnosis add-on therapy
Other: LP with standard of care — The LP will be carried out according to the usual techniques without hypnosis.
  Standard analgesic treatments will be used (except contraindications):
  * EMLA (Lidocain+Prilocain) Cream/Patch
  * Local anesthesia with lidocain chlorhydrate monohydrate 1% injectable
  * Nitrous oxide
  Arms: Lumbar puncture with standard of care

SUMMARY:
The purpose of this study is to assess the effect of hypnosis, as add on therapy, on patients requiring a lumbar puncture (LP) as part of their medical management.

DETAILED DESCRIPTION:
This study will follow the zelen's methodology randomization. It is an add-on study design.

1. The study will be presented to patients as an assessment of their comfort during the LP. The intervention group is not presented to the patient.
2. Patients are asked to sign the consent of the standard of care group.
3. Randomization into two equally sized groups:

   * Intervention arm : LP with complementary hypnoanalgesia
   * Control arm : LP without complementary hypnoanalgesia
4. Patients who have been randomized into the control group, will have LP according to the standard of care.

Patients who have been randomized into the hypnoanalgesic group will be informed about the hypnoanalgesia intervention and then asked to sign the consent of the hypnosis group.

* if the patient accepts, he will benefit from hypnosis during LP.
* if the patient refuses, he will re-join the control group without hypnosis.

The physicians performing LP will be the same in both groups. A phone call follow-up is scheduled on day 3 and 7 after intervention.

ELIGIBILITY:
Inclusion Criteria:

* Required a lumbar puncture for diagnosis
* Affiliated with social security system
* Patient's written consent

Exclusion Criteria:

* LP contraindication
* History of previous LP
* Psychiatric disorder making the realization of a hypnosis irrelevant
* Cognitive-behavioural abilities that do not allow the completion of the study
* Persons who are protected under the act. Person deprived of liberty by judicial decision
* Pregnant or Breastfeeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2021-11-09 (Actual); Primary Completion 2024-03-13 (Actual); Study Completion 2024-03-13 (Actual)

PRIMARY OUTCOMES:
Maximum pain felt during LP | Immediately at the end of LP procedure
  The maximum pain experienced will be assessed in the immediate post procedure using a Numeric Pain Rating Scale (NPRS). The NPRS is a 10 points scale, ranging from 0 (no pain) to 10 (maximal pain).

SECONDARY OUTCOMES:
Comfort felt during LP | Immediately at the end of LP procedure
  The comfort level felt during the LP procedure will be assessed with a Numeric Rating Scale (NRS). The NRS is a 10 points scale, ranging from 0 (total uncomfort) to 10 (maximal comfort).
Ratio of patients with a Numeric Pain Rating Scale (NPRS) score >= 4. | Immediately at the end of LP procedure
  Comparison between the two groups of the ratio of patient with a NPRS >= 4.
Acceptation of hypnosis | Day1
  Number and percentage of subjects randomized and analyzed in the hypnoanalgesia group and who have actually had hypnosis
State and Trait anxiety before LP | Before randomization
  The state and trait anxiety will be assess using the State and Trait anxiety inventory (STAI) questionnaire.
Assess pain at Day 3 and Day 7 | Three days and then seven days after the LP.
  The pain level will be assess using the NPRS scale by telephonic interview.
Timeframe for resumption of usual activities. | Seven days after the LP.
  Number of days between LP and the resumption of usual activities

CONTACTS AND LOCATIONS:
Locations (1):
- Neurology department of Grenoble University Hospital, Grenoble, Isere, France